CLINICAL TRIAL: NCT02534701
Title: ERic Acute StrokE Recanalization (ERASER)
Acronym: ERASER
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: ERASER
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Ischemic Stroke
Keywords: stroke; clot retrieval system; recanalization
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ERIC® and SOFIA™: ERIC® device in combination with SOFIA™ Distal Access Catheter
  Interventions: Device: ERIC® and SOFIA™

INTERVENTIONS:
Device: ERIC® and SOFIA™ — a self-expanding clot retrieval system

SUMMARY:
To monitor the effect of the ERIC® device in combination with SOFIA™ Distal Access Catheter on artery recanalization and on clinical outcomes in stroke patients using data from clinical routine application (ERASER).

To additionally evaluate the effect of the ERIC® device in combination with SOFIA™ Distal Access Catheter on the final infarct volume as determined by advanced image postprocessing methods in the subgroup of patients with acute middle cerebral artery stroke (ERASER+).

DETAILED DESCRIPTION:
This is a prospective, international, single-arm, controlled, open label post-market, multicenter study to compare the safety and effectiveness of ERIC® device in combination with SOFIA™ Distal Access Catheter in acute ischemic stroke patients using clinical routine data.

Patients who meet the imaging inclusion criteria for ERASER will be included in the cohort where collected and additionally analyzed data will be compared to a historical patient cohort (referred to as ERASER imaging =ERASER+). All other patients will be included in a registry (referred to as ERASER), where clinical information will be collected. The overall study duration is expected to be 18 Months. The expected duration of each subject's enrolment is approximately 90 days. Subjects will be followed with assessments at 90 days post stroke.

The basic concept of ERASER+ is the use an infarct prediction algorithm that has been trained on a large dataset of historical imaging data of patients treated with IV tPA, apply it to the pre-treatment imaging and compare its predictions with the actual outcome.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke with NIH-SS score of 8-25
* CTP/ MRP <4.5h after symptom onset completed
* CTA/ MRA confirms M1-occlusion
* Groin puncture estimated <6h after stroke onset
* Intended usage of ERIC® as first device in combination with SOFIA™ Distal Access -Catheter (secondary bail-out with other devices allowed)

Exclusion Criteria:

* MCA >1/3 abnormal in DWI or CBV (ASPECTS ≤ 7, >100 mL)
* Pre stroke mRS ≥ 2
* Necessity of ipsilateral internal carotid artery (ICA) angioplasty
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 year with acute ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
VOST (volume of saved tissue) = VPIv- VMT | 30 h
  volume of saved tissue (VOST) as difference of the brain volume with an infarct risk of >50%, based on a prediction- algorithm trained in a historical cohort treated with IV tPA (VPIv) and the actual infarct volume

SECONDARY OUTCOMES:
mRS≤2 | 90 days
  neurological outcomes (mRS≤2)
NIHSS score improvement ≥10 from baseline | 90 days
  neurological outcomes (NIHSS score improvement ≥10 from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Fiehler, MD,PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (9):
- Germany (8):
  - Universitätsklinikum Augsburg, Augsburg
  - Klinikum Dortmund, Dortmund
  - Universität Greifswald, Greifswald
  - Asklepios Klinik Altona, Hamburg
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Klinikum der Universität München, München
- Kantonspital Aarau, Aarau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fiehler J, Thomalla G, Bernhardt M, Kniep H, Berlis A, Dorn F, Eckert B, Kemmling A, Langner S, Remonda L, Reith W, Rohde S, Mohlenbruch M, Bendszus M, Forkert ND, Gellissen S. ERASER. Stroke. 2019 May;50(5):1275-1278. doi: 10.1161/STROKEAHA.119.024858. PMID 31009356